CLINICAL TRIAL: NCT06239688
Title: Evaluating a National Person-Centered Training Program to Strengthen the Dementia Care Workforce
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-1643; R01AG079124 (NIH)
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Aging; Knowledge, Attitudes, Practice; Long-Term Care; Dementia
Keywords: Workplace Training
MeSH Terms: conditions — Behavior; Dementia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- essentiALZ (Experimental): Communities randomized to this arm will receive the essentiALZ training: a web-based training taken by AL staff that contains three hours of self-paced content separated into five modules, plus a final review. Modules include: 1) Alzheimer's disease and dementia; 2) person-centered care; 3) assessment and care planning; 4) activities of daily living; and 5) behaviors and communication. Staff will be encouraged to take the training over the course of four weeks.
  Interventions: Behavioral: essentiALZ
- essentiALZ + ECHO (Experimental): Communities randomized to this arm will receive the essentiALZ training: a web-based training taken by AL staff that contains three hours of self-paced content separated into five modules, plus a final review. Modules include: 1) Alzheimer's disease and dementia; 2) person-centered care; 3) assessment and care planning; 4) activities of daily living; and 5) behaviors and communication. Staff will be encouraged to take the training over the course of four weeks. Additionally, they will receive access to Project ECHO. ECHO is a virtual tele-mentoring model grounded in case-based learning. It includes six weekly one-hour sessions of didactic and discussive learning. The first five sessions will reflect the content of the five essentiALZ modules, and the final session will address maintenance. ECHO sessions are group sessions that will be conducted via Zoom.
  Interventions: Behavioral: essentiALZ; Behavioral: Project ECHO
- No Intervention (No Intervention): Standard care will be provided.

INTERVENTIONS:
Behavioral: essentiALZ — essentiALZ is a web-based training that contains three hours of self-paced content separated into five modules, plus a final review. Modules include: 1) Alzheimer's disease and dementia; 2) person-centered care; 3) assessment and care planning; 4) activities of daily living; and 5) behaviors and communication. Staff will be encouraged to take the training over the course of four weeks.
  Arms: essentiALZ; essentiALZ + ECHO
Behavioral: Project ECHO — ECHO is a virtual tele-mentoring model grounded in case-based learning. It includes six weekly one-hour sessions of didactic and discussive learning. The first five sessions will reflect the content of the five essentiALZ modules, and the final session will address maintenance. ECHO sessions are group sessions that will be conducted via Zoom.
  Arms: essentiALZ + ECHO

SUMMARY:
This project will compare two training models of an evidence-based online dementia care training program for direct care staff in assisted living to a waitlist control: 1) essentiALZ training and 2) essentiALZ training + Project ECHO. It will examine the extent to which each model is implemented and achieves its intended outcomes to improve staff knowledge and attitudes, change care practices, and improve the wellbeing of staff, residents, and residents' family members. Results will inform next steps in dementia care training for the assisted living (AL) and broader long-term care workforce.

To examine these outcomes, data will be collected from AL staff and families over the course of 6 months. Staff will complete questionnaires and participate in interviews (as applicable) at baseline, post-training, 3-months, and 6-months. Families will participate in interviews at baseline, 3-months, and 6-months.

DETAILED DESCRIPTION:
More than 75% of persons living with Alzheimer's disease and related dementias who reach 80 years of age require residential long-term care, which is increasingly provided in assisted living (AL). Across the country, almost 29,000 AL communities with more than 996,000 beds have become the primary residential care provider for persons with dementia: 90% of AL residents have cognitive impairment and 42% have recorded moderate or severe dementia, with actual rates being higher. AL provides supportive but not nursing services; consequently, virtually all care is provided by direct care workers (nursing assistants and personal care aides).

Unfortunately, direct care workers are undervalued and under-trained, leading to poor care, workplace injury, dissatisfaction, and high turnover. AL is state-regulated, and only 17 states stipulate minimum training hours (some being as low as one hour), meaning that two-thirds of states are silent on training. Fewer than 40% of staff have education beyond high school, and so it is not surprising that a minority report sufficient knowledge to care for persons with dementia. In striving to fill this gap, training for direct care workers must be accessible and have efficacy in benefitting the staff, organization, and persons with dementia.

Online training is an especially promising option due to its low cost, wide availability, and potential for self pacing, automated skills tests, and certification. The Alzheimer's Association is the national leader in dementia care training, and in 2021 developed essentiALZ (pronounced "essentials"), an online program teaching evidence-based, person-centered care, which can be accessed from a computer, tablet, or mobile device. Already more than 1,500 staff have essentiALZ certification, but as is true of the majority of training programs, evidence as to its ability to improve care and outcomes is lacking. It is possible that essentiALZ is effective in changing care and outcomes, but it may also be that additional supports are necessary to do so. A timely model of support is Project ECHO, which has flooded the field of long-term care as a proven way to provide expert guidance and peer support via a remote, online approach. Adding ECHO to online dementia training might provide a necessary boost to achieve care change and improved outcomes.

The project responds to the National Institute on Aging Notice of Special Interest that calls for strengthening the workforce through enhancing and supporting skills training. It will conduct a hybrid implementation/effectiveness randomized trial in 126 AL communities, comparing essentiALZ alone, essentiALZ + ECHO enhancement, and a waitlist control. Outcomes grounded in the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) model and the Kirkpatrick training effectiveness model will be examined over six months, comparing the arms in terms of (1) implementation and (2) effectiveness, and (3) examining the extent to which implementation and effectiveness differ based on characteristics of the AL community, staff, residents, and family members. Results will inform next steps in dementia care training for the AL and broader long-term care workforce.

ELIGIBILITY:
Inclusion Criteria:

AL Staff:

* Staff (part-time, full-time, and including contract staff) who provide direct care to residents at the participating assisted living community (e.g., certified nursing assistants, personal care aides, registered nurses, licensed practical nurses, activity directors, social workers, and others) as determined by the administrator/health care supervisor
* Are 18 years of age or older
* Are able to read and speak English fluently

Family:

* Resident not expected to die or be transferred in the next six months at baseline
* At follow-up, resident lived in AL community at least one month during the three months prior to interview date
* Are a family member/legally authorized representative (LAR), or designated contact of a resident with Alzheimer's disease and related dementia (ADRD) of a participating AL community
* Are 18 years of age or older
* Are English speaking
* Visit the resident at least monthly

Exclusion Criteria:

AL Staff & Family:

- Are under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1764 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Score Over Time of Sense of Competence in Dementia Care (SCIDS) | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  Sense of Competence in Dementia Care (SCIDS) is a 17-item instrument. Responses are indicated using a 4-point Likert scale. Minimum score (worst value) = 1. Maximum score (best value) = 4. Higher values represent a better outcome (range 17-68). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.
Change in Score Over Time of Staff Experience of Working with Residents with Dementia Questionnaire - Care Organization, Satisfactory Contact with the Patient, and Satisfaction with the Expectations of Others Subscales (SEWDRQ) | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  Staff Experience of Working with Residents with Dementia Questionnaire - Care Organization, Satisfactory Contact with the Patient, and Satisfaction with the Expectations of Others Subscales (SEWDRQ) is a 9-item instrument. Responses are indicated using a 5-point Likert scale. Minimum score (worst value) = 0. Maximum score (best value) = 4. Higher values represent a better outcome (range 0-36). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.
Change in Score Over Time of Dementia Attitude Scale - Short Form (DAS-6) | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  Dementia Attitudes Scale (Short-Form) is a 6-item instrument. Responses are indicated using a 7-point Likert scale. Minimum score (worst value) = 1. Maximum score (best value) = 7. Higher values represent a better outcome (range 6-42). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.

SECONDARY OUTCOMES:
Change in Score Over Time of essentiALZ exam items | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  essentiALZ exam items is a 5-item instrument. Instrument is a measure of knowledge on the subject of the intervention training. Responses are multiple choice, with only one answer per question considered 'correct'. Higher values of correct responses represent a better outcome/retention of knowledge (range 0-5). Measure is assessed at Baseline Questionnaire, Post-Training Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.
Change in Score Over Time of essentiALZ organizational practices | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  essentiALZ exam items is a 5-item instrument. Instrument is a measure of knowledge on the subject of the intervention training. Responses are multiple choice, with only one answer per question considered 'correct'. Higher values of correct responses represent a better outcome/retention of knowledge (range 0-5). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.
Change in Score Over Time of Emotional Burnout | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  The researchers will assess intent to leave job by asking "Overall, based on your definition of burnout, how would you rate your level of burnout? Select one." Response options are: "1 = I enjoy my work. I have no symptoms of burnout.", "2 = Occasionally I am under stress, and I don't always have as much energy as I once did, but I don't feel burned out.", "3 - I am definitely burning out and have one or more symptoms of burnout, such as physical and emotional exhaustion.", "4 = The symptoms of burnout that I'm experiencing won't go away. I think about frustration at work a lot.", "5 = I feel completely burned out and often wonder if I can go on. I am at the point where I may need some changes or may need to seek some sort of help." Minimum = 1 (best value), maximum = 5 (worst value). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.
Change in Score Over Time of Intention to Leave | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  The researchers will assess intent to leave job by asking "How likely is it that you will leave this job in the next year? "Would you say... 1 is Not at All Likely, 2 is Somewhat Likely, 3 is Very Likely." Minimum = 1 (best value), maximum = 3 (worst value). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.
Change in Score Over Time of Feeling Valued | Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
  essentiALZ exam items is a 5-item instrument. Instrument is a measure of knowledge on the subject of the intervention training. Responses are multiple choice, with only one answer per question considered 'correct'. Higher values of correct responses represent a better outcome/retention of knowledge (range 0-5). Measure is assessed at Baseline Questionnaire, a 3-month Follow Up Questionnaire and at a 6-month Follow Up Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Zimmerman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified computerized dataset will be available for the use of other researchers. The de-identification of the dataset will follow IRB guidance. Select data will be transformed as appropriate (e.g., items in a scale that were reverse coded will be transformed), and scales will be developed from individual items where indicated (maintaining the individual items).
  The de-identified dataset will be shared in excel or CSV format and will include a codebook for use. Similarly, all data collection instruments will be made available. No specialized tools or software will be necessary to access or use the data. The project coordinator and/or senior analyst will work with potential users for procedures to share the dataset using secure methods informed by Cecil G. Sheps Center for Health Services Data Analytics and Information Technology Department.
Time Frame: A de-identified computerized dataset of all information will be available for the use of other researchers no later than the date of acceptance of the publication that reports the main findings derived from the project, and will remain available for the following ten years.
Access Criteria: Those who wish to use these data will be asked to enter into a data-sharing agreement that will specify the protection of data confidentiality, as well as prohibit the recipient from transferring the data to other users or using the data for purposes other than those expressly agreed upon. In addition, researchers who proposes to use the data will be required to have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable.

REFERENCES:
- [Background] Alzheimer's Disease International. Dementia: A Public Health Priority. Geneva, Switzerland: World Health Organization; 2015.
- [Background] Alzheimer's Association. Alzheimer's Impact Movement March 2018. Costs of Alzheimer's to Medicare and Medicaid. http://act.alz.org/site/DocServer/2012_Costs_Fact_Sheet_version_2.pdf?docID=7161. Accessed October 30, 2021.
- [Background] Langa KM, Larson EB, Crimmins EM, Faul JD, Levine DA, Kabeto MU, Weir DR. A Comparison of the Prevalence of Dementia in the United States in 2000 and 2012. JAMA Intern Med. 2017 Jan 1;177(1):51-58. doi: 10.1001/jamainternmed.2016.6807. PMID 27893041
- [Background] Friedman EM, Shih RA, Langa KM, Hurd MD. US Prevalence And Predictors Of Informal Caregiving For Dementia. Health Aff (Millwood). 2015 Oct;34(10):1637-41. doi: 10.1377/hlthaff.2015.0510. PMID 26438738
- [Background] Arrighi HM, Neumann PJ, Lieberburg IM, Townsend RJ. Lethality of Alzheimer disease and its impact on nursing home placement. Alzheimer Dis Assoc Disord. 2010 Jan-Mar;24(1):90-5. doi: 10.1097/WAD.0b013e31819fe7d1. PMID 19568155
- [Background] Zimmerman S, Gruber-Baldini AL, Sloane PD, Eckert JK, Hebel JR, Morgan LA, Stearns SC, Wildfire J, Magaziner J, Chen C, Konrad TR. Assisted living and nursing homes: apples and oranges? Gerontologist. 2003 Apr;43 Spec No 2:107-17. doi: 10.1093/geront/43.suppl_2.107. PMID 12711731
- [Background] Zimmerman S, Love K, Cohen LW, Pinkowitz J, Nyrop KA. Person-Centeredness in Home- and Community-Based Services and Supports: Domains, Attributes, and Assisted Living Indicators. Clin Gerontol. 2014;37(5):429-445. doi: 10.1080/07317115.2014.937548. Epub 2014 Jun 30. PMID 29033493
- [Background] Smith M, Buckwalter KC, Kang H, Ellingrod V, Schultz SK. Dementia care in assisted living: needs and challenges. Issues Ment Health Nurs. 2008 Aug;29(8):817-38. doi: 10.1080/01612840802182839. PMID 18649209
- [Background] Harris-Kojetin L, Sengupta M, Park-Lee E, Valverde R, Caffrey C, Rome V, Lendon J. Long-Term Care Providers and services users in the United States: data from the National Study of Long-Term Care Providers, 2013-2014. Vital Health Stat 3. 2016 Feb;(38):x-xii; 1-105. PMID 27023287
- [Background] Harrington C, Chapman S, Miller E, et al. Trends in the supply of long-term-care facilities and beds in the United States. J Appl Gerontol 2005;24(4):265-282.
- [Background] Paraprofessional Healthcare Institute. Caring for the Future: The Power and Potential of America's Direct Care Workforce. 2021. http://phinational.org/resource/caring-for-the-future-the-power-andpotential-of-americas-direct-care-workforce/. Accessed October 30, 2021.
- [Background] Han K, Trinkoff AM, Storr CL, Lerner N, Yang BK. Variation Across U.S. Assisted Living Facilities: Admissions, Resident Care Needs, and Staffing. J Nurs Scholarsh. 2017 Jan;49(1):24-32. doi: 10.1111/jnu.12262. Epub 2016 Nov 10. PMID 27860170
- [Background] Zimmerman S, Sloane PD, Williams CS, Dobbs D, Ellajosyula R, Braaten A, Rupnow MF, Kaufer DI. Residential care/assisted living staff may detect undiagnosed dementia using the minimum data set cognition scale. J Am Geriatr Soc. 2007 Sep;55(9):1349-55. doi: 10.1111/j.1532-5415.2007.01289.x. PMID 17767676
- [Background] Rosenblatt A, Samus QM, Steele CD, Baker AS, Harper MG, Brandt J, Rabins PV, Lyketsos CG. The Maryland Assisted Living Study: prevalence, recognition, and treatment of dementia and other psychiatric disorders in the assisted living population of central Maryland. J Am Geriatr Soc. 2004 Oct;52(10):1618-25. doi: 10.1111/j.1532-5415.2004.52452.x. PMID 15450036
- [Background] National Center for Assisted Living. Assisted Living: A Growing Aspect of Long-Term Care. https://www.ahcancal.org/Advocacy/IssueBriefs/NCAL_Factsheet_2019.pdf. Accessed October 30, 2021.
- [Background] Hawes C, Phillips CD, Rose M. High service or high privacy assisted living facilities, their residents and staff: Results from a national survey. Washington, DC: U.S. Department of Health and Human Services; 2000.
- [Background] National Center for Assisted Living (NCAL). 2019. 2019 Assisted Living State Regulatory Review. Washington, DC: NCAL. https://www.ahcancal.org/ncal/advocacy/regs/Documents/2019_reg_review.pdf. Accessed October 30, 2021.
- [Background] Zimmerman S, Williams CS, Reed PS, Boustani M, Preisser JS, Heck E, Sloane PD. Attitudes, stress, and satisfaction of staff who care for residents with dementia. Gerontologist. 2005 Oct;45 Spec No 1(1):96-105. doi: 10.1093/geront/45.suppl_1.96. PMID 16230756
- [Background] Sloane PD, Yearby R, Konetzka RT, Li Y, Espinoza R, Zimmerman S. Addressing Systemic Racism in Nursing Homes: A Time for Action. J Am Med Dir Assoc. 2021 Apr;22(4):886-892. doi: 10.1016/j.jamda.2021.02.023. Epub 2021 Mar 26. PMID 33775548
- [Background] U.S. Department of Health and Human Services. (2013). National Plan to Address Alzheimer's Disease: 2013 Update. http://aspe.hhs.gov/daltcp/napa/ NatlPlan2013.shtml. Accessed October 30, 2021.
- [Background] Scales K, Zimmerman S, Miller SJ. Evidence-Based Nonpharmacological Practices to Address Behavioral and Psychological Symptoms of Dementia. Gerontologist. 2018 Jan 18;58(suppl_1):S88-S102. doi: 10.1093/geront/gnx167. PMID 29361069
- [Background] Beer JM, McBride SE, Mitzner TL, Rogers WA. Understanding challenges in the front lines of home health care: a human-systems approach. Appl Ergon. 2014 Nov;45(6):1687-99. doi: 10.1016/j.apergo.2014.05.019. Epub 2014 Jun 21. PMID 24958610
- [Background] Gould E, Reed P. Alzheimer's Association Quality Care Campaign and professional training initiatives: improving hands-on care for people with dementia in the U.S.A. Int Psychogeriatr. 2009 Apr;21 Suppl 1:S25-33. doi: 10.1017/S1041610209008758. Epub 2009 Mar 17. PMID 19288968
- [Background] Thomas KS, Cornell PY, Zhang W, Smith L, Hua C, Kaskie B, Carder P. The Relationship Between States' Staffing Regulations And Hospitalizations Of Assisted Living Residents. Health Aff (Millwood). 2021 Sep;40(9):1377-1385. doi: 10.1377/hlthaff.2021.00598. PMID 34495716
- [Background] Zimmerman S, Love K, Sloane PD, Cohen LW, Reed D, Carder PC; Center for Excellence in Assisted Living-University of North Carolina Collaborative. Medication administration errors in assisted living: scope, characteristics, and the importance of staff training. J Am Geriatr Soc. 2011 Jun;59(6):1060-8. doi: 10.1111/j.1532-5415.2011.03430.x. Epub 2011 Jun 7. PMID 21649628
- [Background] Castle NG, Engberg J, Mendeloff J, Burns R. A national view of workplace injuries in nursing homes. Health Care Manage Rev. 2009 Jan-Mar;34(1):92-103. doi: 10.1097/01.HMR.0000342981.37673.74. PMID 19104267
- [Background] Campbell S. 2018. Workplace Injuries and the Direct Care Workforce. Bronx, NY: PHI. https://phinational.org/wp-content/ uploads/2018/04/Workplace-Injuries-and-DCW-PHI-2018.pdf. Accessed October 30, 2021.
- [Background] Franzosa E, Tsui EK, Baron S. "Who's Caring for Us?": Understanding and Addressing the Effects of Emotional Labor on Home Health Aides' Well-being. Gerontologist. 2019 Nov 16;59(6):1055-1064. doi: 10.1093/geront/gny099. PMID 30124808
- [Background] Stacey CL. Finding dignity in dirty work: the constraints and rewards of low-wage home care labour. Sociol Health Illn. 2005 Sep;27(6):831-54. doi: 10.1111/j.1467-9566.2005.00476.x. PMID 16283901
- [Background] Edberg AK, Bird M, Richards DA, Woods R, Keeley P, Davis-Quarrell V. Strain in nursing care of people with dementia: nurses' experience in Australia, Sweden and United Kingdom. Aging Ment Health. 2008 Mar;12(2):236-43. doi: 10.1080/13607860701616374. PMID 18389404
- [Background] American Health Care Association. 2012. American Health Care Association 2012 Staffing Report.Washington, DC: AHCA. https://www.ahcancal.org/research_data/staffing/Documents/2012_Staffing_Report.pdf. Accessed October 30, 2021.
- [Background] Hawes C, Rose M, Phillips CD. 1999. A national study of assisted living for the frail elderly: results of a national survey of facilities. Washington, DC: U.S. Department of Health and Human Services, Office of Disability, Aging, and Long-Term Care Policy.
- [Background] Konetzka RT, Stearns SC, Konrad TR, et al. Personal care aide turnover in residential care settings: An assessment of ownership, economic, and environmental factors. J of Appl Gerontol 2005;24(2):87-107.
- [Background] Khatutsky G, Wiener J, Anderson W, et al. 2011. Understanding Direct Care Workers: A Snapshot of Two of America's Most Important Jobs: Certified Nursing Assistants and Home Health Aides. Washington, DC: U.S. Department of Health and Human Services. http://aspe.hhs.gov/daltcp/reports/2011/cnachart.pdf. Accessed October 30, 2021.
- [Background] Seavey D. (2004). The cost of frontline turnover in long-term care. Washington, DC: American Association of Homes and Services for the Aging. https://phinational.org/wpcontent/uploads/legacy/clearinghouse/TOCostReport.pdf. Accessed October 30, 2021.
- [Background] Castle NG, Engberg J, Anderson R, Men A. Job satisfaction of nurse aides in nursing homes: intent to leave and turnover. Gerontologist. 2007 Apr;47(2):193-204. doi: 10.1093/geront/47.2.193. PMID 17440124
- [Background] Dawson SL, Surpin R. Direct-care health workers: you get what you pay for. Generations 2001;25:23-28.
- [Background] Trinkoff AM, Storr CL, Lerner NB, Yang BK, Han K. CNA Training Requirements and Resident Care Outcomes in Nursing Homes. Gerontologist. 2017 Jun 1;57(3):501-508. doi: 10.1093/geront/gnw049. PMID 27059825
- [Background] Kelly CM, Morgan JC, Jason KJ. Home care workers: interstate differences in training requirements and their implications for quality. J Appl Gerontol. 2013 Oct;32(7):804-32. doi: 10.1177/0733464812437371. Epub 2012 Mar 22. PMID 25474799
- [Background] Ahn R. HCIA Complex/High-Risk Patient Targeting: Third Annual Report. 2017. Bethesda, MD: NORC at the University of Chicago. https:// downloads.cms.gov/files/cmmi/hcia-chspt-thirdannualrpt.pdf. Accessed October 30, 2021.
- [Background] McKenzie GL, Teri L, Salazar MK, Farran CJ, Beck C, Paun O. Relationship between system-level characteristics of assisted living facilities and the health and safety of unlicensed staff. AAOHN J. 2011 Apr;59(4):173-80. doi: 10.3928/08910162-20110328-01. PMID 21462900
- [Background] Yeatts DE, Cready C, Swan J, Shen Y. The perception of "training availability" among certified nurse aides: relationship to CNA performance, turnover, attitudes, burnout, and empowerment. Gerontol Geriatr Educ. 2010;31(2):115-32. doi: 10.1080/02701961003795722. PMID 20509059
- [Background] Hollinger-Smith L, Ortigara A. A LEAP toward culture change. Provider. 2006 Feb;32(2):35-8. No abstract available. PMID 16910190
- [Background] Connolly C, Christman A. Surveying the Home Care Workforce: Their Challenges & the Positive Impact of Unionization. 2017. New York, NY: NELP. https://www.nelp.org/publication/surveying-the-home-careworkforce/. Accessed October 30, 2021.
- [Background] Luz CC, Hanson KV, Hao Y, Spurgeon E. Improving Patient Experiences and Outcomes Through Personal Care Aide Training. J Patient Exp. 2018 Mar;5(1):56-62. doi: 10.1177/2374373517724349. Epub 2017 Aug 30. PMID 29582012
- [Background] Surr CA, Parveen S, Smith SJ, Drury M, Sass C, Burden S, Oyebode J. The barriers and facilitators to implementing dementia education and training in health and social care services: a mixed-methods study. BMC Health Serv Res. 2020 Jun 5;20(1):512. doi: 10.1186/s12913-020-05382-4. PMID 32503536
- [Background] Stone R. Introduction: the role of training and education in solving the direct care workforce crisis. Gerontol Geriatr Educ. 2007;28(2):5-16. doi: 10.1300/J021v28n02_02. No abstract available. PMID 18032188
- [Background] Fazio S, Zimmerman S, Doyle PJ, Shubeck E, Carpenter M, Coram P, Klinger JH, Jackson L, Pace D, Kallmyer B, Pike J; members of the Alzheimer's Association Dementia Care Provider Roundtable. What Is Really Needed to Provide Effective, Person-Centered Care for Behavioral Expressions of Dementia? Guidance from The Alzheimer's Association Dementia Care Provider Roundtable. J Am Med Dir Assoc. 2020 Nov;21(11):1582-1586.e1. doi: 10.1016/j.jamda.2020.05.017. Epub 2020 Jul 25. PMID 32723533
- [Background] Kim SK, Park M. Effectiveness of person-centered care on people with dementia: a systematic review and meta-analysis. Clin Interv Aging. 2017 Feb 17;12:381-397. doi: 10.2147/CIA.S117637. eCollection 2017. PMID 28255234
- [Background] Scholzel-Dorenbos CJ, Meeuwsen EJ, Olde Rikkert MG. Integrating unmet needs into dementia health-related quality of life research and care: Introduction of the Hierarchy Model of Needs in Dementia. Aging Ment Health. 2010 Jan;14(1):113-9. doi: 10.1080/13607860903046495. PMID 20155528
- [Background] Pioneer Network. Person-centered care and the new conditions of participation: It's about doing it right! October 24, 2017. https://www.pioneernetwork.net/person-centered-care-new-conditions-participationright/. Accessed October 30, 2021.
- [Background] American Health Care Association/National Center for Assisted Living. https://www.ahcancal.org/Assisted-Living/Pages/default.aspx. Accessed October 30, 2021.
- [Background] Sloane PD, Hoeffer B, Mitchell CM, McKenzie DA, Barrick AL, Rader J, Stewart BJ, Talerico KA, Rasin JH, Zink RC, Koch GG. Effect of person-centered showering and the towel bath on bathing-associated aggression, agitation, and discomfort in nursing home residents with dementia: a randomized, controlled trial. J Am Geriatr Soc. 2004 Nov;52(11):1795-804. doi: 10.1111/j.1532-5415.2004.52501.x. PMID 15507054
- [Background] Zimmerman S, Sloane PD, Ward K, Wretman CJ, Stearns SC, Poole P, Preisser JS. Effectiveness of a Mouth Care Program Provided by Nursing Home Staff vs Standard Care on Reducing Pneumonia Incidence: A Cluster Randomized Trial. JAMA Netw Open. 2020 Jun 1;3(6):e204321. doi: 10.1001/jamanetworkopen.2020.4321. PMID 32558913
- [Background] Ballard C, Corbett A, Orrell M, Williams G, Moniz-Cook E, Romeo R, Woods B, Garrod L, Testad I, Woodward-Carlton B, Wenborn J, Knapp M, Fossey J. Impact of person-centred care training and person-centred activities on quality of life, agitation, and antipsychotic use in people with dementia living in nursing homes: A cluster-randomised controlled trial. PLoS Med. 2018 Feb 6;15(2):e1002500. doi: 10.1371/journal.pmed.1002500. eCollection 2018 Feb. PMID 29408901
- [Background] Ordway A, Johnson KL, Kneale L, Amtmann D, Demiris G. The Experience of Home Care Providers and Beneficiaries With Enhanced Training Requirements in Washington State. J Aging Health. 2019 Dec;31(10_suppl):124S-144S. doi: 10.1177/0898264319860298. Epub 2019 Jul 3. PMID 31267811
- [Background] Peterson D, Berg-Weger MS, McGillick J, Schwartz L. Basic care I: the effect of dementia-specific training on certified nursing assistants and other staff. Am J Alzheimers Dis Other Demen. 2002 May-Jun;17(3):154-64. doi: 10.1177/153331750201700309. PMID 12083345
- [Background] Polacsek M, Goh A, Malta S, Hallam B, Gahan L, Cooper C, Low LF, Livingston G, Panayiotou A, Loi S, Omori M, Savvas S, Batchelor F, Ames D, Doyle C, Scherer S, Dow B. 'I know they are not trained in dementia': Addressing the need for specialist dementia training for home care workers. Health Soc Care Community. 2020 Mar;28(2):475-484. doi: 10.1111/hsc.12880. Epub 2019 Oct 23. PMID 31646701
- [Background] Reblin M, Uchino BN. Social and emotional support and its implication for health. Curr Opin Psychiatry. 2008 Mar;21(2):201-5. doi: 10.1097/YCO.0b013e3282f3ad89. PMID 18332671
- [Background] Person-Centred dementia care. Making services better Dawn Brooker Person-Centred Dementia Care. Making Services Better Jessica Kingsley 160 pound14.99 1 84310 337 0 1843103370 [Formula: see text]. Nurs Older People. 2007 Jun 1;19(5):22-23. doi: 10.7748/nop.19.5.22.s21. PMID 27726617
- [Background] Kitwood T. Dementia reconsidered: the person comes first. Buckingham, England: Open University Press; 1997.
- [Background] Choi J, Kim DE, Yoon JY. Person-Centered Care Environment Associated With Care Staff Outcomes in Long-Term Care Facilities. J Nurs Res. 2020 Nov 30;29(1):e133. doi: 10.1097/JNR.0000000000000412. PMID 33252502
- [Background] Brownie S, Nancarrow S. Effects of person-centered care on residents and staff in aged-care facilities: a systematic review. Clin Interv Aging. 2013;8:1-10. doi: 10.2147/CIA.S38589. Epub 2013 Jan 3. PMID 23319855
- [Background] Barbosa A, Sousa L, Nolan M, Figueiredo D. Effects of Person-Centered Care Approaches to Dementia Care on Staff: A Systematic Review. Am J Alzheimers Dis Other Demen. 2015 Dec;30(8):713-22. doi: 10.1177/1533317513520213. PMID 24449039
- [Background] Barbosa A, Nolan M, Sousa L, Figueiredo D. Supporting direct care workers in dementia care: effects of a psychoeducational intervention. Am J Alzheimers Dis Other Demen. 2015 Mar;30(2):130-8. doi: 10.1177/1533317514550331. Epub 2014 Sep 18. PMID 25237132
- [Background] Fazio S, Pace D, Maslow K, Zimmerman S, Kallmyer B. Alzheimer's Association Dementia Care Practice Recommendations. Gerontologist. 2018 Jan 18;58(suppl_1):S1-S9. doi: 10.1093/geront/gnx182. No abstract available. PMID 29361074
- [Background] Dobbs D, Hobday J, Roker R, Kaas MJ, Molinari V. Certified nursing assistants' perspectives of the CARES(R) activities of daily living dementia care program. Appl Nurs Res. 2018 Feb;39:244-248. doi: 10.1016/j.apnr.2017.11.016. Epub 2017 Nov 7. PMID 29422166
- [Background] Williams KN, Coleman CK, Perkhounkova Y, Beachy T, Hein M, Shaw CA, Berkley A. Moving Online: A Pilot Clinical Trial of the Changing Talk Online Communication Education for Nursing Home Staff. Gerontologist. 2021 Nov 15;61(8):1338-1345. doi: 10.1093/geront/gnaa210. PMID 33346349
- [Background] Egan KJ, Pinto-Bruno AC, Bighelli I, Berg-Weger M, van Straten A, Albanese E, Pot AM. Online Training and Support Programs Designed to Improve Mental Health and Reduce Burden Among Caregivers of People With Dementia: A Systematic Review. J Am Med Dir Assoc. 2018 Mar;19(3):200-206.e1. doi: 10.1016/j.jamda.2017.10.023. Epub 2018 Jan 4. PMID 29306605
- [Background] Fletcher A, Zimmerman S. Preisser JS, et al. Implementation fidelity of a standardized dementia care training program across multiple trainers and settings. Alz Care Today 2010;11(1):51-60.
- [Background] Pleasant M, Molinari V, Dobbs D, Meng H, Hyer K. Effectiveness of online dementia caregivers training programs: A systematic review. Geriatr Nurs. 2020 Nov-Dec;41(6):921-935. doi: 10.1016/j.gerinurse.2020.07.004. Epub 2020 Jul 20. PMID 32703628
- [Background] Irvine AB, Billow MB, Bourgeois M, Seeley JR. Mental illness training for long term care staff. J Am Med Dir Assoc. 2012 Jan;13(1):81.e7-13. doi: 10.1016/j.jamda.2011.01.015. Epub 2011 Mar 22. PMID 21450251
- [Background] Rosen J, Mulsant BH, Kollar M, Kastango KB, Mazumdar S, Fox D. Mental health training for nursing home staff using computer-based interactive video: a 6-month randomized trial. J Am Med Dir Assoc. 2002 Sep-Oct;3(5):291-6. doi: 10.1097/01.JAM.0000027201.90817.21. PMID 12807615
- [Background] Hattink B, Meiland F, van der Roest H, Kevern P, Abiuso F, Bengtsson J, Giuliano A, Duca A, Sanders J, Basnett F, Nugent C, Kingston P, Droes RM. Web-Based STAR E-Learning Course Increases Empathy and Understanding in Dementia Caregivers: Results from a Randomized Controlled Trial in the Netherlands and the United Kingdom. J Med Internet Res. 2015 Oct 30;17(10):e241. doi: 10.2196/jmir.4025. PMID 26519106
- [Background] Irvine AB, Bourgeois M, Billow M, Seeley JR. Internet training for nurse aides to prevent resident aggression. J Am Med Dir Assoc. 2007 Oct;8(8):519-26. doi: 10.1016/j.jamda.2007.05.002. PMID 17931576
- [Background] Irvine AB, Billow MB, Gates DM, Fitzwater EL, Seeley JR, Bourgeois M. Internet training to respond to aggressive resident behaviors. Gerontologist. 2012 Feb;52(1):13-23. doi: 10.1093/geront/gnr069. Epub 2011 Oct 30. PMID 22038338
- [Background] Su HF, Koo M, Lee WL, Sung HC, Lee RP, Liu WI. A dementia care training using mobile e-learning with mentoring support for home care workers: a controlled study. BMC Geriatr. 2021 Feb 16;21(1):126. doi: 10.1186/s12877-021-02075-3. PMID 33593287
- [Background] Pleasant ML, Molinari V, Hobday JV, Fazio S, Cullen N, Hyer K. An evaluation of the CARES(R) Dementia Basics Program among caregivers. Int Psychogeriatr. 2017 Jan;29(1):45-56. doi: 10.1017/S1041610216001526. Epub 2016 Oct 3. PMID 27692028
- [Background] Bryan JL, Asghar-Ali AA. Development and Dissemination of an Interprofessional Online Dementia Training Curriculum. J Am Geriatr Soc. 2020 Jan;68(1):192-197. doi: 10.1111/jgs.16240. Epub 2019 Nov 6. PMID 31693177
- [Background] Gkioka M, Teichmann B, Moraitou D, Papagiannopoulos S, Tsolaki M. Effects of a Person Centered Dementia Training Program in Greek Hospital Staff-Implementation and Evaluation. Brain Sci. 2020 Dec 12;10(12):976. doi: 10.3390/brainsci10120976. PMID 33322754
- [Background] Surr CA, Gates C, Irving D, Oyebode J, Smith SJ, Parveen S, Drury M, Dennison A. Effective Dementia Education and Training for the Health and Social Care Workforce: A Systematic Review of the Literature. Rev Educ Res. 2017 Oct;87(5):966-1002. doi: 10.3102/0034654317723305. Epub 2017 Jul 31. PMID 28989194
- [Background] Miller HV, Ward K, Zimmerman S. Implementation effectiveness of psychosocial and environmental care practices in assisted living. Geriatr Nurs. 2021 Jan-Feb;42(1):295-302. doi: 10.1016/j.gerinurse.2020.09.003. Epub 2020 Oct 8. PMID 33041084
- [Background] Ploeg J, Skelly J, Rowan M, Edwards N, Davies B, Grinspun D, Bajnok I, Downey A. The role of nursing best practice champions in diffusing practice guidelines: a mixed methods study. Worldviews Evid Based Nurs. 2010 Dec;7(4):238-51. doi: 10.1111/j.1741-6787.2010.00202.x. Epub 2010 Sep 28. PMID 20880009
- [Background] Drake A. How 'upskilling' can maximize home care workers' contributions and improve serious illness care. Health Affairs Blog. 2019. DOI: 10.1377/hblog20190227.420595. Accessed October 30, 2021.
- [Background] Arora S, Geppert CM, Kalishman S, Dion D, Pullara F, Bjeletich B, Simpson G, Alverson DC, Moore LB, Kuhl D, Scaletti JV. Academic health center management of chronic diseases through knowledge networks: Project ECHO. Acad Med. 2007 Feb;82(2):154-60. doi: 10.1097/ACM.0b013e31802d8f68. PMID 17264693
- [Background] Cuttriss N, Bouchonville MF, Maahs DM, Walker AF. Tele-rounds and Case-Based Training: Project ECHO Telementoring Model Applied to Complex Diabetes Care. Pediatr Clin North Am. 2020 Aug;67(4):759-772. doi: 10.1016/j.pcl.2020.04.017. Epub 2020 Jun 19. PMID 32650871
- [Background] Thies KM, Gonzalez M, Porto A, Ashley KL, Korman S, Lamb M. Project ECHO COVID-19: Vulnerable Populations and Telehealth Early in the Pandemic. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211019286. doi: 10.1177/21501327211019286. PMID 34036832
- [Background] Arora S, Thornton K, Murata G, Deming P, Kalishman S, Dion D, Parish B, Burke T, Pak W, Dunkelberg J, Kistin M, Brown J, Jenkusky S, Komaromy M, Qualls C. Outcomes of treatment for hepatitis C virus infection by primary care providers. N Engl J Med. 2011 Jun 9;364(23):2199-207. doi: 10.1056/NEJMoa1009370. Epub 2011 Jun 1. PMID 21631316
- [Background] Baughman AW, Renton M, Wehbi NK, Sheehan EJ, Gregorio TM, Yurkofsky M, Levine S, Jackson V, Pu CT, Lipsitz LA. Building community and resilience in Massachusetts nursing homes during the COVID-19 pandemic. J Am Geriatr Soc. 2021 Oct;69(10):2716-2721. doi: 10.1111/jgs.17389. Epub 2021 Aug 3. PMID 34310686
- [Background] Zimmerman S, Gould E, Reed PS, Sloane PD. Dementia care training in nursing homes and assisted living: part I. Alz Care Today 2010;11(1).
- [Background] Zimmerman S, Gould E, Reed PS, Sloane PD. Dementia care training in nursing homes and assisted living: part II. Alz Care Today 2010;11(2).
- [Background] Fletcher A, Zimmerman S. Preisser JS, et al. Trainee and trainer reactions to a scripted dementia care training program in residential care/assisted living settings and nursing homes. Alz Care Today 2010;11(1):61-70.
- [Background] McConnell ES, Corazzini KN, Lekan D, et al. Perception of new pain care practices in dementia care: psychometric properties of the Duke Diffusion of Innovation in Long-Term Care Battery. Alz Care Today 2010;11(2):122-133.
- [Background] Mitchell CM, Zimmerman S, Beeber AS. Dementia care training in long-term care: if you provide it, will they come? Alz Care Today 2010:11(1):40-50.
- [Background] Zimmerman S, Mitchell CM, Reed D, et al. Outcomes of a dementia care training program for staff in nursing homes and residential care/assisted living settings. Alz Care Today 2010;11(2):83-99.
- [Background] Corazzini KN, McConnell ES, Anderson RA, et al. The importance of organizational climate to training needs and outcomes in long-term care. Alz Care Today 2010;11(2):109-121.
- [Background] Bates R. A critical analysis of evaluation practice: The Kirkpatrick model and the principle of beneficence. Eval Program Plann 2004;27:341-347.
- [Background] Kirkpatrick D. Techniques for evaluating training programs. Train Dev J 1979;33(6):79-92.
- [Background] Brody AA, Galvin JE. A review of interprofessional dissemination and education interventions for recognizing and managing dementia. Gerontol Geriatr Educ. 2013;34(3):225-56. doi: 10.1080/02701960.2013.801342. PMID 23879387
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Holtrop JS, Estabrooks PA, Gaglio B, Harden SM, Kessler RS, King DK, Kwan BM, Ory MG, Rabin BA, Shelton RC, Glasgow RE. Understanding and applying the RE-AIM framework: Clarifications and resources. J Clin Transl Sci. 2021 May 14;5(1):e126. doi: 10.1017/cts.2021.789. eCollection 2021. PMID 34367671
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658
- [Background] Carder PC. State Regulatory Approaches for Dementia Care in Residential Care and Assisted Living. Gerontologist. 2017 Aug 1;57(4):776-786. doi: 10.1093/geront/gnw197. PMID 28077453
- [Background] U.S. Department of Health and Human Services. Compendium of Residential Care and Assisted Living Regulations and Policy: 2015 Edition. https://aspe.hhs.gov/sites/default/files/migrated_legacy_files//73501/15alcom.pdf. Accessed October 30, 2021.
- [Background] US Census Bureau. https://www.census.gov/quickfacts/fact/table/US/PST045219. Accessed October 30, 2021.
- [Background] Zimmerman S, Sloane PD, Eckert JK, Gruber-Baldini AL, Morgan LA, Hebel JR, Magaziner J, Stearns SC, Chen CK. How good is assisted living? Findings and implications from an outcomes study. J Gerontol B Psychol Sci Soc Sci. 2005 Jul;60(4):S195-204. doi: 10.1093/geronb/60.4.s195. PMID 15980295
- [Background] Hawes C, Phillips CD, Rose M, Holan S, Sherman M. A national survey of assisted living facilities. Gerontologist. 2003 Dec;43(6):875-82. doi: 10.1093/geront/43.6.875. PMID 14704387
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. Milbank Q. 2004;82(4):581-629. doi: 10.1111/j.0887-378X.2004.00325.x. PMID 15595944
- [Background] Cho H, ed. Health Communication Message Design: Theory and Practice. Thousand Oaks, CA: SAGE Publications; 2012.
- [Background] Doak CC, Doak LG, Root JH. Teaching Patients with Low Literacy Skills, 2nd Ed. Philadelphia: Lippincott Williams & Wilkins; 1995.
- [Background] Plain Language Action and Information Network. Plain language in healthcare. https://plainlanguage.gov/resources/content-types/healthcare/. Accessed October 30, 2021.
- [Background] Houts PS, Doak CC, Doak LG, Loscalzo MJ. The role of pictures in improving health communication: a review of research on attention, comprehension, recall, and adherence. Patient Educ Couns. 2006 May;61(2):173-90. doi: 10.1016/j.pec.2005.05.004. Epub 2005 Aug 24. PMID 16122896
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Zimmerman S, Greene A, Sloane PD, Mitchell M, Giuliani C, Nyrop K, Walsh E. Preventing falls in assisted living: Results of a quality improvement pilot study. Geriatr Nurs. 2017 May-Jun;38(3):185-191. doi: 10.1016/j.gerinurse.2016.09.003. Epub 2016 Oct 21. PMID 27776786
- [Background] Sloane PD, Zimmerman S, Ward K, Kistler CE, Paone D, Weber DJ, Wretman CJ, Preisser JS. A 2-Year Pragmatic Trial of Antibiotic Stewardship in 27 Community Nursing Homes. J Am Geriatr Soc. 2020 Jan;68(1):46-54. doi: 10.1111/jgs.16059. Epub 2019 Jul 18. PMID 31317534
- [Background] Harris-Wallace B, Schumacher JG, Perez R, Eckert JK, Doyle PJ, Beeber AS, Zimmerman S. The Emerging Role of Health Care Supervisors in Assisted Living. Seniors Hous Care J. 2011 Jan 1;19(1):97-108. PMID 24817991
- [Background] Port CL, Zimmerman S, Williams CS, Dobbs D, Preisser JS, Williams SW. Families filling the gap: comparing family involvement for assisted living and nursing home residents with dementia. Gerontologist. 2005 Oct;45 Spec No 1(1):87-95. doi: 10.1093/geront/45.suppl_1.87. PMID 16230755
- [Background] Cohen LW, Zimmerman S, Reed D, Sloane PD, Beeber AS, Washington T, Cagle JG, Gwyther LP. Dementia in relation to family caregiver involvement and burden in long-term care. J Appl Gerontol. 2014 Aug;33(5):522-40. doi: 10.1177/0733464813505701. Epub 2013 Oct 16. PMID 24652906
- [Background] Schneider J, Schonstein A, Teschauer W, Kruse A, Teichmann B. Hospital Staff's Attitudes Toward and Knowledge About Dementia Before and After a Two-Day Dementia Training Program. J Alzheimers Dis. 2020;77(1):355-365. doi: 10.3233/JAD-200268. PMID 32741821
- [Background] Sloane PD, Williams CS, Zimmerman S. Immigrant status and intention to leave of nursing assistants in U.S. nursing homes. J Am Geriatr Soc. 2010 Apr;58(4):731-7. doi: 10.1111/j.1532-5415.2010.02781.x. PMID 20398155
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Zimmerman S, Hawkes WG, Hebel JR, Fox KM, Lydick E, Magaziner J. The Lower Extremity Gain Scale: a performance-based measure to assess recovery after hip fracture. Arch Phys Med Rehabil. 2006 Mar;87(3):430-6. doi: 10.1016/j.apmr.2005.10.026. PMID 16500180
- [Background] Munn JC, Dobbs D, Meier A, Williams CS, Biola H, Zimmerman S. The end-of-life experience in long-term care: five themes identified from focus groups with residents, family members, and staff. Gerontologist. 2008 Aug;48(4):485-94. doi: 10.1093/geront/48.4.485. PMID 18728298
- [Background] Lydick E, Zimmerman SI, Yawn B, Love B, Kleerekoper M, Ross P, Martin A, Holmes R. Development and validation of a discriminative quality of life questionnaire for osteoporosis (the OPTQoL). J Bone Miner Res. 1997 Mar;12(3):456-63. doi: 10.1359/jbmr.1997.12.3.456. PMID 9076589
- [Background] Project ECHO Evaluation 101: A Practical Guide for Evaluating Your Program. https://nyshealthfoundation.org/wp-content/uploads/2017/12/project-echo-evaluation-guide.pdf. Accessed October 30, 2021.
- [Background] Lintern T,Woods B, Phair L. Training is not enough to change care practice. J Demen Care 2000;8:15-17.
- [Background] Surr CA, Smith SJ, Crossland J, Robins J. Impact of a person-centred dementia care training programme on hospital staff attitudes, role efficacy and perceptions of caring for people with dementia: A repeated measures study. Int J Nurs Stud. 2016 Jan;53:144-51. doi: 10.1016/j.ijnurstu.2015.09.009. Epub 2015 Sep 25. PMID 26421910
- [Background] de Vries K, Drury-Ruddlesden J, McGill G. Investigation into attitudes towards older people with dementia in acute hospital using the Approaches to Dementia Questionnaire. Dementia (London). 2020 Nov;19(8):2761-2779. doi: 10.1177/1471301219857577. Epub 2019 Jun 21. PMID 31226896
- [Background] Schepers AK, Orrell M, Shanahan N, Spector A. Sense of competence in dementia care staff (SCIDS) scale: development, reliability, and validity. Int Psychogeriatr. 2012 Jul;24(7):1153-62. doi: 10.1017/S104161021100247X. Epub 2012 Feb 20. PMID 22340666
- [Background] Banks P, Waugh A, Henderson J, Sharp B, Brown M, Oliver J, Marland G. Enriching the care of patients with dementia in acute settings? The Dementia Champions Programme in Scotland. Dementia (London). 2014 Nov;13(6):717-36. doi: 10.1177/1471301213485084. Epub 2013 May 1. PMID 24339079
- [Background] Nakanishi M, Endo K, Hirooka K, Nakashima T, Morimoto Y, Granvik E, Minthon L, Nagga K, Nishida A. Dementia behaviour management programme at home: impact of a palliative care approach on care managers and professional caregivers of home care services. Aging Ment Health. 2018 Aug;22(8):1057-1062. doi: 10.1080/13607863.2017.1332160. Epub 2017 May 29. PMID 28553880
- [Background] Astrom S, Nilsson M, Norberg A, Sandman PO, Winblad B. Staff burnout in dementia care--relations to empathy and attitudes. Int J Nurs Stud. 1991;28(1):65-75. doi: 10.1016/0020-7489(91)90051-4. PMID 1856035
- [Background] National Nursing Assistant Questionnaire, 2006. https://www.cdc.gov/nchs/data/nnhsd/2004NNASQuestionnaire.pdf. Accessed October 30, 2021.
- [Background] Moyle W, Murfield JE, Griffiths SG, Venturato L. Care staff attitudes and experiences of working with older people with dementia. Australas J Ageing. 2011 Dec;30(4):186-90. doi: 10.1111/j.1741-6612.2010.00470.x. Epub 2010 Oct 8. PMID 22176562
- [Background] Dolan ED, Mohr D, Lempa M, Joos S, Fihn SD, Nelson KM, Helfrich CD. Using a single item to measure burnout in primary care staff: a psychometric evaluation. J Gen Intern Med. 2015 May;30(5):582-7. doi: 10.1007/s11606-014-3112-6. Epub 2014 Dec 2. PMID 25451989
- [Background] Zimmerman S, Cohen LW, Reed D, Gwyther LP, Washington T, Cagle JG, Sloane PD, Preisser JS. Families Matter in Long-Term Care: Results of a Group-Randomized Trial. Seniors Hous Care J. 2013;21(1):3-20. PMID 25243051
- [Background] Maas ML, Reed D, Park M, Specht JP, Schutte D, Kelley LS, Swanson EA, Trip-Reimer T, Buckwalte KC. Outcomes of family involvement in care intervention for caregivers of individuals with dementia. Nurs Res. 2004 Mar-Apr;53(2):76-86. doi: 10.1097/00006199-200403000-00003. PMID 15084992
- [Background] Donner A, Klar N. Design and analysis of cluster randomization trials in health research. Arnold: London, 2000.
- [Background] Sloane PD, Zimmerman S, Perez R, Reed D, Harris-Wallace B, Khandelwal C, Beeber AS, Mitchell CM, Schumacher J. Physician perspectives on medical care delivery in assisted living. J Am Geriatr Soc. 2011 Dec;59(12):2326-31. doi: 10.1111/j.1532-5415.2011.03714.x. Epub 2011 Nov 8. PMID 22091932
- [Background] Zimmerman S, Dobbs D, Roth EG, Goldman S, Peeples AD, Wallace B. Promoting and Protecting Against Stigma in Assisted Living and Nursing Homes. Gerontologist. 2016 Jun;56(3):535-47. doi: 10.1093/geront/gnu058. Epub 2014 Jun 13. PMID 24928555
- [Background] Morgan LA, Eckert JK, Gruber-Baldini AL, Zimmerman S. Policy and research issues for small assisted living facilities. J Aging Soc Policy. 2004;16(4):1-16. doi: 10.1300/J031v16n04_01. PMID 15724570
- [Background] Dobbs D, Zimmerman S, Carder P, Beeber AS, Palmertree SJ. Staff Reports of Behavioral Expressions of Persons With Dementia in 250 Assisted Living Communities. Gerontologist. 2022 Feb 9;62(2):169-180. doi: 10.1093/geront/gnab059. PMID 33993241
- [Background] van Soest-Poortvliet MC, van der Steen JT, Zimmerman S, Cohen LW, Munn J, Achterberg WP, Ribbe MW, de Vet HC. Measuring the quality of dying and quality of care when dying in long-term care settings: a qualitative content analysis of available instruments. J Pain Symptom Manage. 2011 Dec;42(6):852-63. doi: 10.1016/j.jpainsymman.2011.02.018. Epub 2011 May 26. PMID 21620642
- [Background] Kistler CE, Sloane PD, Platts-Mills TF, Beeber AS, Khandelwal C, Weber DJ, Mitchell CM, Reed D, Chisholm L, Zimmerman S. Challenges of antibiotic prescribing for assisted living residents: perspectives of providers, staff, residents, and family members. J Am Geriatr Soc. 2013 Apr;61(4):565-70. doi: 10.1111/jgs.12159. Epub 2013 Mar 1. PMID 23452167
- [Background] Schumacher JG, Eckert JK, Zimmerman S, Carder P, Wright A. Physician care in assisted living: a qualitative study. J Am Med Dir Assoc. 2005 Jan-Feb;6(1):34-45. doi: 10.1016/j.jamda.2004.12.005. PMID 15871869
- [Background] Green J, Thorogood N. Qualitative Methods for Health Research. 2nd Ed. Los Angeles: SAGE; 2009.
- [Background] Glaser BG, Strauss AL. The Discovery of Grounded Theory. Chicago, IL: Aldine; 1967.
- [Background] Hooper R, Teerenstra S, de Hoop E, Eldridge S. Sample size calculation for stepped wedge and other longitudinal cluster randomised trials. Stat Med. 2016 Nov 20;35(26):4718-4728. doi: 10.1002/sim.7028. Epub 2016 Jun 28. PMID 27350420
- [Background] Li F, Turner EL, Preisser JS. Optimal allocation of clusters in cohort stepped wedge designs. Statistics and Probability Letters 2018; 137:257-263.